CLINICAL TRIAL: NCT06179407
Title: A Two-Part Study to Assess the Safety, Tolerability, Pharmacokinetics and Sleep Latency Effects of MK-6552 in Participants With Narcolepsy Type 1
Brief Title: Study of MK-6552 in Participants With Narcolepsy Type 1 (MK-6552-004)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated for business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 6552-004; MK-6554-004 (Other: MSD)
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-6552 (Experimental): In Part 1, participants will receive single oral doses of MK-6552 in ascending fashion approximately 6 hours apart for a single day, based on safety and tolerability of the previous dose. In Part 2, participants will receive multiple days of MK-6552 dosing (7 consecutive days) at the highest safe and well tolerated MK-6552 dose determined on an individual basis from Part 1.
  Interventions: Drug: MK-6552
- Placebo (Placebo Comparator): In Part 2, participants will receive multiple days of placebo dosing (7 consecutive days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-6552 — Oral capsule administered according to allocation (Part 1)/randomization (Part 2).
  Arms: MK-6552
Drug: Placebo — In Part 2, participants will receive multiple days of placebo dosing (7 consecutive days).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of MK-6552 in participants with Narcolepsy Type 1 (NT1). Part 1 will evaluate safety, tolerability, and PK of MK-6552 after administration of ascending doses in a single day to support a dose level decision for Part 2. Part 2 will investigate the PD of MK-6552 after single-day and multiple-day administration. Participants who complete Part 1 and demonstrate that they are able to tolerate at least one dose level of MK-6552 will participate in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of NT1, including a valid polysomnography within the previous 5 years and a current diagnosis of NT1 for at least 6 months based on criteria established by the International Classification of Sleep Disorders- Third Edition, or Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) [American Psychiatric Association 2013]
* Is positive for HLA-DQB1*06:02 allele supporting a diagnosis of NT1
* Has a baseline history of unequivocal cataplexy prior to initiation of anti-cataplexy medications
* Reports a total sleep time of > 6 hours on at least 4 out of 7 nights each week within the 4 weeks prior to screening visit

Exclusion Criteria:

* Has history of or current hypertension
* Has underlying cardiovascular or cerebrovascular conditions in which an acute rise in blood pressure would pose a clinical concern, including but nor limited to aneurysms or arteriovenous malformations
* Has a history of renal or hepatic impairment
* Has a history of cardiac ischemia or cerebral ischemia including but not limited to history of stroke, transient ischemic attack, or transient global amnesia
* Based on clinical interview and responses on the Columbia-Suicide Severity Rating Scale, is at imminent risk of self-harm or of harm to others in the opinion of the investigator
* Mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years
* History of cancer (malignancy)
* Has a history of any of the following sleep disorders: obstructive sleep apnea (OSA) defined as an Apnea Hypopnea Index > 15 per hour per the American Academy of Sleep Medicine alternate criteria, primary insomnia (within the past 6 months), circadian rhythm sleep disorder, shift work sleep disorder (within the past 6 months), clinically significant parasomnia at the discretion of the investigator
* Has a history of seizure disorder, clinically significant head trauma, or past invasive intracranial surgery or clinically significant dementia
* Positive test(s) for Hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing an Adverse Event (AE) | Up to approximately 9 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that experience an AE will be reported.
Number of participants discontinuing study intervention due to an Adverse Event (AE) | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants that discontinue study intervention due to an AE will be reported.
Sleep Onset Latency Measured by the Maintenance of Wakefulness Test (MWT) | 1 hour after each dose on Day 7
  The MWT is a daytime polysomnographic procedure that measures objectively the ability to remain awake during sleep-inducing circumstances. Sleep onset latency is defined as the first occurrence of sustained sleep (i.e. 3 consecutive 30 second epochs of N1 [stage 1] sleep or any single 30 second epoch of N2 [stage 2], N3 [stage 3 and 4 combined] or REM). The primary outcome measure of sleep onset latency measured by the MWT on Day 7 will be reported.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve of MK-6552 from Time Zero to infinity (AUC0-inf) | Day 1 Dose 1: Predose, 0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose 1. Day 1 Dose 2: 0.25, 0.5, 1, 2, 3, 4, 6, 8, 18, 21 and 24 hours postdose
  Blood samples will be collected at specified intervals for the determination of AUC0-inf. AUC0-inf is defined as the area under the concentration-time curve of MK-6552 from time zero to infinity and will be reported for participants in Part 1.
Area Under the Plasma Concentration-Time Curve of MK-6552 from Time Zero to 24 hours postdose (AUC0-24) | Day 1 Dose 1: Predose, 0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose 1. Day 1 Dose 2: 0.25, 0.5, 1, 2, 3, 4, 6, 8, 18, 21 and 24 hours postdose
  Blood samples will be collected at specified intervals for the determination of AUC0-24. AUC0-24 is defined as the area under the concentration-time curve of MK-6552 from time zero to 24 hours postdose and will be reported for participants in Part 1.
Time to Maximum Concentration (Tmax) of MK-6552 | Day 1 Dose 1: Predose, 0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose 1. Day 1 Dose 2: 0.25, 0.5, 1, 2, 3, 4, 6, 8, 18, 21 and 24 hours postdose
  Blood samples will be collected at specified intervals for the determination of Tmax. Tmax is defined as the time to the maximum concentration of MK-6552 reached and will be reported for participants in Part 1.
Maximum Concentration (Cmax) of MK-6552 | Day 1 Dose 1: Predose, 0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose 1. Day 1 Dose 2: 0.25, 0.5, 1, 2, 3, 4, 6, 8, 18, 21 and 24 hours postdose
  Blood samples will be collected at specified intervals for the determination of Cmax. Cmax is defined as the maximum concentration of MK-6552 reached and will be reported for participants in Part 1.
Concentration of MK-6522 at 2 Hours Postdose (C2h) | Day 1: 2 hours postdose
  Blood samples will be collected at specified intervals for the determination of C2h. C2h is defined as the concentration of MK-6552 reached at 2 hours postdose and will be reported for participants in Part 1.
Concentration of MK-6522 at 6 Hours Postdose (C6h) | Day 1: 6 hours post Dose 1
  Blood samples will be collected at specified intervals for the determination of C6h. C6h is defined as the concentration of MK-6552 reached at 6 hours post Dose 1 and will be reported for participants in Part 1.
Concentration of MK-6522 at 18 Hours Postdose (C18h) | 18 hours post Day 1 Dose 2
  Blood samples will be collected at specified intervals for the determination of C18h. C18h is defined as the concentration of MK-6552 reached at 18 hours post Dose 2 and will be reported for participants in Part 1.
Apparent Oral Clearance (CL/F) of MK-6552 | Day 1 Dose 1: Predose, 0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose 1. Day 1 Dose 2: 0.25, 0.5, 1, 2, 3, 4, 6, 8, 18, 21 and 24 hours postdose
  Blood samples will be collected at specified intervals for the determination of CL/F. CL/F is defined as the rate at which MK-6552 is completely removed from plasma and will be reported for participants in Part 1.
Apparent Volume of Distribution (Vz/F) of MK-6552 | Day 1 Dose 1: Predose, 0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose 1. Day 1 Dose 2: 0.25, 0.5, 1, 2, 3, 4, 6, 8, 18, 21 and 24 hours postdose
  Blood samples will be collected at specified intervals for the determination of Vz/F. Vz/F is defined as the theoretical volume that would be necessary to contain the total amount of administered MK-6522 at the same concentration that it is observed in the blood plasma, and will be reported for participants in Part 1.
Apparent Terminal Half-life (t½) of MK-6552 | Day 1 Dose 1: Predose, 0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose 1. Day 1 Dose 2: 0.25, 0.5, 1, 2, 3, 4, 6, 8, 18, 21 and 24 hours postdose
  Blood samples will be collected at specified intervals for the determination of t½. t½ is defined as the time required to divide the MK-6552 plasma concentration by two after reaching pseudo-equilibrium, and will be reported for participants in Part 1.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- United States (5):
  - Delta Waves, Inc. ( Site 0008), Colorado Springs, Colorado
  - Teradan Clinical Trials, LLC ( Site 0005), Brandon, Florida
  - NeuroTrials Research Inc ( Site 0006), Atlanta, Georgia
  - Bogan Sleep Consultants ( Site 0001), Columbia, South Carolina
  - FutureSearch Trials of Neurology ( Site 0004), Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com